CLINICAL TRIAL: NCT01278186
Title: Prospective Randomized Study of the Paclitaxel-Coated Balloon Catheter in Bifurcated Coronary Lesions / BABILON Study (Paclitaxel-Coated Balloon in Bifurcated Lesions)
Brief Title: Study of the Paclitaxel-Coated Balloon Catheter in Bifurcated Coronary Lesions
Acronym: BABILON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: B.Braun Surgical SA (Industry)
Collaborators: Hospital Universitario Infanta Cristina de Badajoz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-0909
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary stenosis; Bifurcation; Drug-eluting balloon; Drug-eluting stent; Angiographic follow-up; Late Lumen Loss; Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Paclitaxel-eluting balloon (Experimental): Paclitaxel-eluting balloon catheter (SeQuent Please, B. Braun)
  Interventions: Procedure: Balloon angioplasty
- Paclitaxel-eluting stent (Experimental): Paclitaxel-eluting stent
  Interventions: Procedure: Stent implantation

INTERVENTIONS:
Procedure: Balloon angioplasty — Coronary angioplasty using the paclitaxel-coated balloon catheter
  Other Names: SeQuent Please
  Arms: Paclitaxel-eluting balloon
Procedure: Stent implantation — Coronary angioplasty using the paclitaxel-eluting stent
  Other Names: Paclitaxel-eluting stent
  Arms: Paclitaxel-eluting stent

SUMMARY:
This study in bifurcated coronary lesions compares the new technology of the paclitaxel-eluting balloon with the usual technique until now of "provisional stenting" with the paclitaxel-eluting stent in the main branch.

DETAILED DESCRIPTION:
The bifurcated coronary lesions are still a challenge for interventional cardiologists, since there is no suitable technique or strategy to manage such lesions.

This multicenter randomized prospective trial in bifurcated coronary lesions will compare the new technology of the paclitaxel-eluting balloon with the until now "gold standard" technique of the "provisional stenting" with the paclitaxel DES in the main branch.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

* Patients with stable angina (1-3) or unstable angina (1-3 A-C) or documented silent ischemia
* Patients with mental and logistic conditions for the follow-up
* Patients should accept an angiographic follow-up at 9 months, a clinical follow-up at 3 years and sign the consent

LESIONS

* De-novo lesions in the bifurcations of DA/Diag either CX/OM or CD/DP with diameters in the main vessel of 2,5 to 3,8/ 2 to 3,5 and lengths < 22 mm
* The left main lesions in bifurcation are also accepted but with another independent randomization list (specify at randomization)
* The diameter of the stenoses should be >50% in any branch with documented ischemia or more than 70% in absence of an ischemia test
* Single vessel or multivessel disease
* In case of a PTCA of more than one lesion, the non included lesion should be treated previously to the included lesion

Exclusion Criteria:

PATIENTS

* Patients with STEMI < 72 hours
* Patients with congestive heart failure or NYHA IV, shock or severe valvular heart disease
* Patients with short life expectancy, or with problems for platelet antiaggregation
* Patients in treatment with hyperthyroidism, in treatment with immunosuppression or anticoagulants, or with alcohol or drug addiction
* Patients included in other trials
* Patients with a stroke 6 months before
* Patients with a surgery one week before
* Severe renal failure calculated as GF < 30 ml/min "Cockcroft Gault"
* Women of childbearing age, with probability to become pregnant during the first year of follow-up

LESIONS

* Evidence of important thrombus within the vessel to treat
* Patients with another stent previously implanted at ≤ 15 mm from the current lesion of the study
* Lesions affecting bypass
* Chronic occlusions to treat
* Restenosis in-stent or of a segment in 4 mm close to the target lesion
* Severe calcification not totally dilatable with the balloon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) | Late angiographic follow-up (9 months)
  Assessment of the difference between both groups regarding the Late Lumen Loss (LLL) in main vessel and side branch, measured at late angiographic follow-up at 9 months
Restenosis | Late angiographic follow-up (9 months)
  Assessment of the difference between both groups regarding the Restenosis in both branches (proximal part of the main vessel, distal part of the main vessel and side branch), measured at late angiographic follow-up at 9 months

SECONDARY OUTCOMES:
Thrombosis rate | Late angiographic follow-up (9 months)
  Assesment of the thrombosis rate
Target Lesion Revascularization (TLR) | Late angiographic follow-up (9 months)
  Assessment of the Target Lesion Revascularization (TLR) at late angiographic follow-up (9 months) if dilatation by restenosis or previous angiography due to angina
Major Adverse Cardiac Events (MACE) | Late angiographic follow-up (9 months)
  Assessment of the rate of Major Adverse Cardiac Events (MACE): death, AMI, Target Lesion Revascularization (TLR) - due to angina pectoris or angiographic restenosis-

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ramon Lopez-Minguez, MD, PhD, Study Director — Hospital Universitario Infanta Cristina de Badajoz
Locations (9):
- Spain (9):
  - Hospital Universitario Infanta Cristina, Badajoz, Badajoz
  - Hospital Universitari Son Dureta, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario San Pedro de Alcantara, Cáceres, Caceres
  - Hospital Universitario Puerta del Mar, Cadiz, Cadiz
  - Hospital Universitario de Puerto Real, Puerto Real, Cadiz
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Virgen de la Salud, Toledo, Toledo

REFERENCES:
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Lefevre T, Louvard Y, Morice MC, Dumas P, Loubeyre C, Benslimane A, Premchand RK, Guillard N, Piechaud JF. Stenting of bifurcation lesions: classification, treatments, and results. Catheter Cardiovasc Interv. 2000 Mar;49(3):274-83. doi: 10.1002/(sici)1522-726x(200003)49:33.0.co;2-n. PMID 10700058
- [Background] Koo BK, Kang HJ, Youn TJ, Chae IH, Choi DJ, Kim HS, Sohn DW, Oh BH, Lee MM, Park YB, Choi YS, Tahk SJ. Physiologic assessment of jailed side branch lesions using fractional flow reserve. J Am Coll Cardiol. 2005 Aug 16;46(4):633-7. doi: 10.1016/j.jacc.2005.04.054. PMID 16098427
- [Background] Yamashita T, Nishida T, Adamian MG, Briguori C, Vaghetti M, Corvaja N, Albiero R, Finci L, Di Mario C, Tobis JM, Colombo A. Bifurcation lesions: two stents versus one stent--immediate and follow-up results. J Am Coll Cardiol. 2000 Apr;35(5):1145-51. doi: 10.1016/s0735-1097(00)00534-9. PMID 10758954
- [Background] Colombo A, Moses JW, Morice MC, Ludwig J, Holmes DR Jr, Spanos V, Louvard Y, Desmedt B, Di Mario C, Leon MB. Randomized study to evaluate sirolimus-eluting stents implanted at coronary bifurcation lesions. Circulation. 2004 Mar 16;109(10):1244-9. doi: 10.1161/01.CIR.0000118474.71662.E3. Epub 2004 Feb 23. PMID 14981005
- [Background] Pan M, de Lezo JS, Medina A, Romero M, Segura J, Pavlovic D, Delgado A, Ojeda S, Melian F, Herrador J, Urena I, Burgos L. Rapamycin-eluting stents for the treatment of bifurcated coronary lesions: a randomized comparison of a simple versus complex strategy. Am Heart J. 2004 Nov;148(5):857-64. doi: 10.1016/j.ahj.2004.05.029. PMID 15523318
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Hildick-Smith D, The BBC ONE (British Bifurcation Coronary study: Old, New and Evolving strategies). Transcatheter Cardiovascular Therapeutics 2008; Oct 12-17. 2008. Washington DC. TCT 2008
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Delgado A, Segura J, Ojeda S, Pavlovic D, Ariza J, Fernandez-Duenas J, Herrador J, Urena I. [Six-month intravascular ultrasound follow-up of coronary bifurcation lesions treated with rapamycin-eluting stents: technical considerations]. Rev Esp Cardiol. 2005 Nov;58(11):1278-86. Spanish. PMID 16324581
- [Background] Suárez de Lezo J, Medina A, Martín P, Amador C, Delgado A, Suárez de Lezo J et al. Hallazgos ultrasónicos durante el tratamiento percutáneo de lesiones coronarias en bifurcaciones. Rev Esp Cardiol 2008;61:930-5
- [Background] Medina A, Suarez de Lezo J, Pan M. [A new classification of coronary bifurcation lesions]. Rev Esp Cardiol. 2006 Feb;59(2):183. No abstract available. Spanish. PMID 16540043
- [Background] Dzavik V, Kharbanda R, Ivanov J, Ing DJ, Bui S, Mackie K, Ramsamujh R, Barolet A, Schwartz L, Seidelin PH. Predictors of long-term outcome after crush stenting of coronary bifurcation lesions: importance of the bifurcation angle. Am Heart J. 2006 Oct;152(4):762-9. doi: 10.1016/j.ahj.2006.04.033. PMID 16996856
- [Background] Ong AT, McFadden EP, Regar E, de Jaegere PP, van Domburg RT, Serruys PW. Late angiographic stent thrombosis (LAST) events with drug-eluting stents. J Am Coll Cardiol. 2005 Jun 21;45(12):2088-92. doi: 10.1016/j.jacc.2005.02.086. PMID 15963413
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Scheller B, Speck U, Schmitt A, Bohm M, Nickenig G. Addition of paclitaxel to contrast media prevents restenosis after coronary stent implantation. J Am Coll Cardiol. 2003 Oct 15;42(8):1415-20. doi: 10.1016/s0735-1097(03)01056-8. PMID 14563585
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Axel DI, Kunert W, Goggelmann C, Oberhoff M, Herdeg C, Kuttner A, Wild DH, Brehm BR, Riessen R, Koveker G, Karsch KR. Paclitaxel inhibits arterial smooth muscle cell proliferation and migration in vitro and in vivo using local drug delivery. Circulation. 1997 Jul 15;96(2):636-45. doi: 10.1161/01.cir.96.2.636. PMID 9244237
- [Background] Posa A, Hemetsberger R, Petnehazy O, Petrasi Z, Testor M, Glogar D, Gyongyosi M. Attainment of local drug delivery with paclitaxel-eluting balloon in porcine coronary arteries. Coron Artery Dis. 2008 Jun;19(4):243-7. doi: 10.1097/MCA.0b013e3283030b26. PMID 18480668
- [Background] Nikol S, Huehns TY, Hofling B. Molecular biology and post-angioplasty restenosis. Atherosclerosis. 1996 Jun;123(1-2):17-31. doi: 10.1016/0021-9150(96)05807-8. No abstract available. PMID 8782834
- [Background] Scheller B. Drug-Eluting Balloons: The B.BRAUN Paclitaxel-Eluting Balloon Program: Device Characteristics, Experimental Findings, and Clinical. Outcomes in Patients with In-Stent Restenosis and for Small Vessels (PEPCAD I and II). Transcatheter Cardiovascular Therapeutics 2008; Oct 12-17
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Additional Ongoing BRAUN Paclitaxel-Eluting Balloon Clinical Trials in Diabetics,Bifurcations and Chronic Total Occlusions (Other PEPCAD Studies). Mathey DG. Transcatheter Cardiovascular Therapeutics 2008;October 12-17, 2008 • Washington, DC.
- [Background] Fanggiday JC, Stella PR, Guyomi SH, Doevendans PA. Safety and efficacy of drug-eluting balloons in percutaneous treatment of bifurcation lesions: the DEBIUT (drug-eluting balloon in bifurcation Utrecht) registry. Catheter Cardiovasc Interv. 2008 Apr 1;71(5):629-35. doi: 10.1002/ccd.21452. PMID 18360855
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Background] Ferrerio JL, Cequier A, Gómez JA, Maristany J, Fernández F, Gómez M et al. Contraindicaciones al inicio o interrupción precoz de la doble antiagregación en pacientes con indicación de intervencionismo coronario percutáneo. Rev Esp Cardiol 2007;60 Supl 2:1-192 pag 149.